CLINICAL TRIAL: NCT05351008
Title: Effects of Cognitive Functional Therapy in Individuals With Chronic Neuropathic Low Back Pain
Brief Title: Effects of CFT in Individuals With CNLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Evgenia Trevlaki, Principal Investigator, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IntHellenicUniv
Record Dates: First submitted 2022-04-07; First posted 2022-04-28 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain; Neuropathic Low Back Pain
Keywords: Chronic pain; Neuropathic pain; Low back pain
MeSH Terms: conditions — Chronic Pain; Neuralgia; Low Back Pain | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Two arms, parallel-design, assessor-blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Functional Therapy group (Experimental): The group will receive 4 months 1 times per week of cognitive functional therapy.
  Interventions: Other: Cognitive Functional Therapy
- Core strengthening group (Active Comparator): The group will receive 4 months 1 times per week of an exercise program aming core strengthening.
  Interventions: Other: Exercise program:

INTERVENTIONS:
Other: Cognitive Functional Therapy — A physicaltheapy approach combining cognitive techniques, func-tional movement training, functional integration and Lifestyle Changes.
  Arms: Cognitive Functional Therapy group
Other: Exercise program: — Core strengthening program
  Arms: Core strengthening group

SUMMARY:
This research aims to deepen the understanding of the interplay between chronic neuropathic low back pain and its effects on physical health, mental well-being, and overall quality of life. Additionally, it will evaluate the impact of cognitive functional therapy (CFT) and core strengthening programs on managing chronic neuropathic low back pain. The study is grounded in the hypothesis that CFT will offer a comprehensive, multidisciplinary, and holistic therapeutic approach for individuals suffering from chronic neuropathic low back pain.

DETAILED DESCRIPTION:
In July 2020, the International Association for the Study of Pain (IASP) revised the definition of pain, according to which pain is an unpleasant aesthetic and emotional experience related to, or appears to be related to, real or potential tissue damage. Chronic pain is characterized by a long duration, exceeding 6 months. Chronic neuropathic pain is caused by damage or disease of the somatosensory nervous system.

Cognitive Functional Therapy (CFT) is a multidimensional, patient-centred intervention that directly explores and manages cognitive, psychological and social factors deemed to be barriers to recovery in chronic low back pain (Vibe Fersum K et al., 2013; Meziat Filho, 2015; Meziat Filho et al., 2016; O'Keeffe et al., 2015a; Rabey et al., 2015; Meziat-Filho et al., 2018). The CFT approach centres on the retraining of maladaptive movement patterns, reconceptualising patient pain beliefs, and addressing any relevant cognitive, psychological, social or lifestyle factors (O'Sullivan P., 2005). CFT is an integrated behavioral approach for individualizing the management of people with disabling LBP once serious (eg, malignancy, infection, inflammatory disorder, and fracture) and specific pathology (eg, nerve root compression with progressive neurological deficit with or without cauda equina symptoms) has been excluded (O'Sullivan et al., 2018).

ELIGIBILITY:
Eligible participants were

* adults (aged ≥18 years) with chronic (≥ 3 months) low back pain prior to surgery,
* who consent and compliance with all aspects of the study protocol, methods, providing data during follow-up contact.

Exclusion criteria were

* serious spinal pathology (eg, fracture, infection, or cancer),
* any medical condition that prevented being physically active,
* being pregnant or having given birth within the previous year,
* inadequate Greek literacy for the study's questionnaires and instructions,
* surgery scheduled within 4 months,
* BMI greater than 40 kg/m2,
* history of psychogenic illness or manic episode,
* history of other neuromuscular disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | through study completion, an average of 2 year
  Short-form McGill Pain Questionnaire (SF-MPQ) is a pain rating index with 2 scales: Sensory subscale with 11 words, and Affective subscale with 4 words from the original MPQ. Minimum value 0, maximum value 5.
Disability | through study completion, an average of 2 years
  Roland-Morris Disability Questionnaire (RDQ), is a 24-item patient-reported outcome measure that inquiries about pain-related disability resulting from low back pain (LBP). The end score is the sum of the ticked boxes. The score ranges from 0 (no disability) to 11, 18 or 24 (max. disability) depending on the questionnaire that is used.

SECONDARY OUTCOMES:
Fear-Avoidance Beliefs | through study completion, an average of 2 years
  Fear-Avoidance Beliefs Questionnaire (FABQ)
Anxiety | through study completion, an average of 2 years
  Generalised Anxiety Disorder Assessment (GAD-7) is a 7-item, self-administered patient questionnaire used as a screening tool and severity measure for generalised anxiety disorder (GAD). A score of 10 or greater on the GAD-7 represents a reasonable cut point for identifying cases of GAD. Cut points of 5, 10, and 15 might be interpreted as representing mild, moderate, and severe levels of anxiety on the GAD-7.
Depression | through study completion, an average of 2 years
  Patient Health Questionnaire-9 (PHQ-9) is a 9-item, self-administered screening instrument for detecting MDD based on the DSM-IV diagnostic criteria. A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Quality of Life as an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. | through study completion, an average of 2 years
  WHO Quality of life - bref is a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment. The measure is calculated by summing the point values for the questions corresponding to each domain and then transforming the scores to a 0-100 point interval, or alternatively, a 4-20 point interval.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra-Hristara Papadopoulou, Professor, Study Chair — International Hellenic University
Locations (1):
- Physical Therapy Clinic Trevlakis Emmanouil, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No